CLINICAL TRIAL: NCT04009018
Title: Adaptation of Perioperative Satisfaction Scale in Regional Anesthesia and Investigation of Its Psychometric Properties
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ömer Faruk Boran (Other)
Responsible Party: Sponsor-Investigator, Ömer Faruk Boran, Clinical Professor, Kahramanmaras Sutcu Imam University
Organization: Kahramanmaras Sutcu Imam University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Regional-1
Record Dates: First submitted 2019-06-26; First posted 2019-07-05 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Scales, Repression-Sensitization; Anesthesia Awareness
Keywords: scale; validity; reliability
MeSH Terms: conditions — Intraoperative Awareness | interventions — Anesthesia, Conduction; Surveys and Questionnaires

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psycometric analyses (Other): It will be a validation study of the Perioperative Satisfaction Scale in Regional Anesthesia. This study is not experimental research. This is a psychometric assessment study of a questionnaire and data will collect pencil-paper survey and face to face from the patients who will get regional anesthesia in the postoperative second day.
  Interventions: Other: Perioperative Satisfaction Scale in Regional Anesthesia

INTERVENTIONS:
Other: Perioperative Satisfaction Scale in Regional Anesthesia — This study is methodological research. Perioperative Satisfaction Scale in Regional Anesthesia will be used to collect data.
  Other Names: Measurement tool (Questionnaire)

SUMMARY:
The aim of the study is to determine the psychometric properties of Perioperative Satisfaction Scale in Regional Anesthesia. In the Turkish version of the scale, a blind reverse translation method will use. And validity and reliability analyses will conduct.

DETAILED DESCRIPTION:
The aim of the present research is to contribute to the international literature determining and describing the factor structure and psychometric qualities of the Perioperative Satisfaction Scale in Regional Anesthesia. An additional aim is to contribute to the national literature regarding the performance of the instrument in cross-cultural adaptation. The following steps will be taken: (a) translation of the scale from English into Turkish, (b) data collection, and (c) checking validity and reliability evidence for the adapted Perioperative Satisfaction Scale in Regional Anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the research
* Participants are over 18 years of age
* Provided regional anesthesia
* Postoperative second day
* No cognitive problems in self-expression

Exclusion Criteria:

* Lack of Turkish literacy
* Use of anesthesia technique other than regional anesthesia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2019-06-20 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction | postoperative 48 hours
  Perioperative Satisfaction Scale in Regional Anesthesia will be applied, side effects such as nausea-vomiting, drowsiness will be noted. Patient satisfaction will be assessed with these methods as bad, medium, good, and very good.

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Mehmet Yazar, MD, Study Chair — Kahramanmaras Sutcu Imam University
Locations (1):
- Kahramanmaras Sutcu Imam University, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mui WC, Chang CM, Cheng KF, Lee TY, Ng KO, Tsao KR, Hwang FM. Development and validation of the questionnaire of satisfaction with perioperative anesthetic care for general and regional anesthesia in Taiwanese patients. Anesthesiology. 2011 May;114(5):1064-75. doi: 10.1097/ALN.0b013e318216e835. PMID 21455058
- [Result] Maurice-Szamburski A, Bruder N, Loundou A, Capdevila X, Auquier P. Development and validation of a perioperative satisfaction questionnaire in regional anesthesia. Anesthesiology. 2013 Jan;118(1):78-87. doi: 10.1097/ALN.0b013e31827469f2. PMID 23221859
- See also: Original validation study of Perioperative Satisfaction Scale in Regional Anesthesia — https://www.ncbi.nlm.nih.gov/pubmed/23221859